CLINICAL TRIAL: NCT00607256
Title: A Multi-center, Long-term, Open-label Study of [S,S]-Reboxetine (PNU-165442G) Administered Once Daily in Patients With Fibromyalgia
Brief Title: Long-term OL Study of [S,S]-RBX in Patients With Fibromyalgia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6061046
Record Dates: First submitted 2008-01-23; First posted 2008-02-05 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — O-methyl reboxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: [S,S]-reboxetine

INTERVENTIONS:
Drug: [S,S]-reboxetine — S_S reboxetine dosed daily.

SUMMARY:
To evaluate the lon-term safety and tolerability of [S,S]-reboxetine in patients with fibromyalgia

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of patients meeting the ACR criteria for fibromyalgia (i.e. widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites)

Exclusion Criteria:

* Patients with other severe pain (e.g. DPN and PHN) that may confound assessment or self-evaluation of the pain associated with fibromyalgia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2007-10-20 (Actual); Primary Completion 2009-05-18 (Actual); Study Completion 2009-05-18 (Actual)

PRIMARY OUTCOMES:
12-lead ECG | 68 weeks
Hematology/Biochemistry | 68 weeks
Adverse events | 68 weeks
Physical examination | 68 weeks
Vital signs | 68 weeks

SECONDARY OUTCOMES:
Patient Global Impression of Change | 68 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (74):
- United States (36):
  - Pfizer Investigational Site, Orangevale, California
  - Pfizer Investigational Site, Santa Ana, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Moline, Illinois
  - Pfizer Investigational Site, Prairie Village, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Jefferson City, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Kenilworth, New Jersey
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Staten Island, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Marion, Ohio
  - Pfizer Investigational Site, Medford, Oregon
  - Pfizer Investigational Site, Bethlehem, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Cranston, Rhode Island
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Lincoln, Rhode Island
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Anderson, South Carolina
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Greer, South Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Lake Jackson, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Belgium (2):
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Pellenberg
- Canada (4):
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Moncton, New Brunswick
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
- Czechia (4):
  - Pfizer Investigational Site, Hlučín
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Zlín
- France (3):
  - Pfizer Investigational Site, Lille, Cedex
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
- Germany (7):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Eichstätt
  - Pfizer Investigational Site, Göppingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Mannheim
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Wiesbaden
- Netherlands (3):
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Emmen
  - Pfizer Investigational Site, Leeuwarden
- South Africa (4):
  - Pfizer Investigational Site, Boksburg, Gauteng
  - Pfizer Investigational Site, Pretoria, Gauteng
  - Pfizer Investigational Site, Panorama, Western Cape
  - Pfizer Investigational Site, Parow, Western Cape
- South Korea (2):
  - Pfizer Investigational Site, Suwon, Kyeongki-do
  - Pfizer Investigational Site, Gwangju
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Stockholm
- United Kingdom (6):
  - Pfizer Investigational Site, Cambridge
  - Pfizer Investigational Site, Colchester
  - Pfizer Investigational Site, Derby
  - Pfizer Investigational Site, Dudley, West Midlands
  - Pfizer Investigational Site, Greenock
  - Pfizer Investigational Site, Paisley

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061046&StudyName=Long-term%20OL%20study%20of%20%5BS%2CS%5D-RBX%20in%20patients%20with%20fibromyalgia